CLINICAL TRIAL: NCT00098098
Title: A Phase 1, Open-Label, Dose-Escalating Study to Evaluate the Safety, Tolerability and Immunogenicity of Recombinant Botulinum Vaccine A/B in Healthy Adults
Brief Title: Study to Evaluate the Safety, Tolerability and Immunogenicity of Recombinant Botulinum Vaccine A/B in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DynPort Vaccine Company LLC, A GDIT Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: rBV A/B-01
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: RECOMBINANT BOTULINUM VACCINE A/B
Keywords: Botulinum; Recombinant Botulinum Vaccine; botulinum neurotoxins

INTERVENTIONS:
Biological: rBV A/B

SUMMARY:
The purpose of this trial is to evaluate the safety and tolerability of a two-dose regimen (Day 0 and Day 28) of recombinant Botulinum Vaccine (rBV) A/B in healthy volunteers when given intramuscularly at three ascending dosage levels by cohort and a two-dose regimen (Day 0 and Day 28) of a formulation containing only antigens at the 40 ug total immunizing protein dosage level.

DETAILED DESCRIPTION:
The Phase 1 clinical trial is designed as a single-center, open-label, non-randomized study to evaluate the safety, tolerability and immunogenicity of a two-dose schedule of rBV A/B in healthy volunteers at three ascending dosage levels, 5 ug, 10 ug and 20 ug serotype-specific antigen (10 ug, 20 ug and 40 ug total immunizing protein) in three dosing cohorts and a two-dose regimen (Day 0 and Day 28) of a formulation containing only antigens at the 40 ug total immunizing protein dosage level. Approximately 44 volunteers (11 per cohort) are expected to be enrolled. Cohorts will enroll consecutively beginning with the lowest dosage level. Volunteers in each cohort will receive a two injection series at the assigned dosage level given as a 0.5 mL intramuscular (i.m.) injection on Day 0 and Day 28. Potential volunteers for study participation will undergo qualification screening for this study during the 21 days prior to the date scheduled for vaccination. After successful completion of the informed consent process and all screening assessments, volunteers will be scheduled for vaccination. Volunteers will report acute adverse events daily for 28 days after each vaccination and return to the clinic at regular intervals according to the Schedule of Study Assessments with the last scheduled follow-up 168 days (± 7 days) after the initial vaccination (Day 0).

ELIGIBILITY:
Inclusion Criteria

* The volunteer is between 18 to 40 (inclusive) years of age at the time of the first dose of rBV A/B.
* The volunteer is in good health as determined by the Investigator (Study Doctor) from a medical history and physical examination.
* The volunteer has clinical chemistry, hematology and urinalysis laboratory values within 10 % above the upper or within 10 % below the lower limit of the normal range as established by the University of Kentucky clinical laboratory which are not considered clinically significant by the Investigator and/or the Sponsor Medical Monitor.
* The volunteer has a normal electrocardiogram (ECG). However, if a potential volunteer is reported to have a benign ECG abnormality (e.g., sinus bradycardia) the results may be discussed with the Sponsor Medical Monitor. With the agreement of the Sponsor Medical Monitor and documentation of the consultation in the volunteer's study record, the Investigator may include the volunteer in the study.
* The volunteer is willing to have his or her blood samples stored for future botulinum research studies.
* The volunteer has signed the Informed Consent Form, successfully completed (at least 90 % correct) the Test of Understanding, and has signed the Health Insurance Portability and Accountability Act (HIPAA) authorization form.
* The volunteer agrees not to donate blood for at least 30 days following vaccination.
* The volunteer is willing to comply with the requirements of the protocol through the post-vaccination Day 168 (± 7 days) visit.
* Female volunteers must be of non-childbearing potential (i.e., surgically sterilized or postmenopausal), or must not be pregnant (as indicated by a negative serum pregnancy test within 24 hours prior to rBV A/B administration) or nursing, and must use two types of acceptable form of FDA-approved birth control methods including: 1) hormonal types of birth control (such as implants or birth control pills) or an intrauterine device (IUD) and 2) an additional barrier type of birth control measure (i.e. condoms, diaphragms, cervical caps, spermicide, etc.) during the period beginning from 30 days before vaccination through completion of the study. Completion of the study is defined as completing the post-vaccination Day 168 (± 7 days) visit.

Exclusion Criteria

* The volunteer has frequent or severe headaches of any etiology.
* The volunteer has chronic, severe or recurrent joint pain or arthritis of any etiology.
* The volunteer has a history of alcohol or drug abuse within the 12 months prior to study screening or any history of injectable drug use.
* The volunteer has a positive result on a urine drug screen that tests for common substances of abuse such as amphetamines, barbiturates, benzodiazepines, cocaine, opiates, and cannabinoids. (If positive on screen, confirmatory testing shall be performed where applicable).
* The volunteer has a previous diagnosis of any serious psychiatric disorder. For this purpose, serious psychiatric disorder is defined as illness requiring hospitalization within the previous 12 months; routine administration of more than one medication to control anxiety, mood or sleep disorder; or history of suicide attempt.
* The volunteer has received any blood products or immune globulin in the previous six months.
* The volunteer has donated blood within the past 56 days.
* The volunteer received any investigational drug therapy within 30 days before the first dose of rBV A/B or intends to receive any other investigational drug therapy before the post-vaccination Day 168 (± 7 days) visit.
* Licensed vaccines are not exclusionary but should be given at least 30 days before or after immunization (if live vaccine: 60 days before or after immunization) to avoid potential confusion of adverse reactions.
* The volunteer has received any other investigational Botulinum Vaccine or Toxoid.
* The volunteer has received previous treatment with approved therapeutic products containing botulinum neurotoxins such as Botox, Myobloc, and Botox Cosmetic.
* The volunteer has a clinically significant abnormality on the ECG.
* The volunteer has a known hypersensitivity to aluminum compounds or yeast.
* The volunteer has any laboratory values greater than 10 % above the upper or greater than 10 % below the lower limit of normal or clinically significant as assessed by the Investigator and/or Sponsor Medical Monitor.
* The volunteer tests positive for Human Immunodeficiency Virus (HIV); Hepatitis C Virus (HCV) or Hepatitis B surface Antigen (HBsAg).
* The volunteer has a body mass index > 40 kg/m2 or is > 100 lbs. over ideal body weight.
* The volunteer has an acute illness, evidence of significant active infection, or evidence of systemic disease at time of enrollment that in the opinion of the Investigator would place the volunteer at an unacceptable risk for injury.
* The volunteer has a temperature > 100.4 °F at the time of enrollment.
* The volunteer has occupational or other responsibilities that would prevent completion of participation in the study.
* The volunteer has a history of anaphylaxis or other serious adverse reactions to vaccines.
* The volunteer has a personal or family history of multiple sclerosis.
* The female volunteer is pregnant (must have a negative serum pregnancy test within 24 hours prior to each dose of rBV A/B), lactating or unwilling to use two types of an acceptable form of FDA-approved contraception for 30 days prior to first dose of rBV A/B through the post-vaccination Day 168 (± 7 days) visit.
* The volunteer requires chemotherapeutic and immunosuppressive agents or a total corticosteroid dose of 2 mg/kg or 20 mg/day within the 3 months prior to the study or burst steroid therapy within 14 days before vaccination.
* The volunteer is currently on active duty in the US military.
* The volunteer is a US military veteran that received other botulinum products for vaccination or research purposes.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2004-08; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of rBV A/B in healthy volunteers at three ascending dosage levels by cohort and a two-dose regimen of a formulation containing only antigens at the 40 ug dosage level.

SECONDARY OUTCOMES:
To evaluate the neutralizing antibody concentration of rBV A/B
Evaluate human toxin neutralizing antibody as a correlate of protective immunity.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greenberg, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States